CLINICAL TRIAL: NCT04871750
Title: Prospective, Randomized Controlled Study on the Effects of Dietary Soy Protein on Facial
Brief Title: Effects of Dietary Soy Protein on Facial Wrinkles in Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: United Soybean Board (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYW_01
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Photoaging
Keywords: Facial Wrinkles; Soy-derived isoflavone; Short-chain fatty acids; Gut microbiome; Dermatology; Supplementation
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: Healthy postmenopausal women aged 50 to 70, with Fitzpatrick skin type I or II.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy protein (Experimental): 30 g powder/day, contains 50 mg of isoflavones
  Interventions: Dietary Supplement: Soy protein
- Casein protein (Placebo Comparator): 30 g powder/day, no isoflavones
  Interventions: Dietary Supplement: Casein protein

INTERVENTIONS:
Dietary Supplement: Soy protein — Daily consumption for 24 weeks
  Arms: Soy protein
Dietary Supplement: Casein protein — Daily consumption for 24 weeks
  Arms: Casein protein

SUMMARY:
Soy and soy-derived products are the primary dietary sources of isoflavones, particularly daidzein and genistein, for humans. Isoflavones are noted to have several effects on the skin including proliferation of keratinocytes resulting in epidermal thickening and increasing collagen and moisture content of the skin. Previous work has shown that the ingestion of an oral supplement containing soy isoflavones as a component led to a clinically measurable improvement in wrinkle depth after 14 weeks of supplementation.

Ingestion of soy-based products has been shown to shift the Bifidobacteria and Lactobacilli among the gut microbiota and modulate the ratio of Firmicutes to Bacteroidetes. Many studies have shown that short-chain fatty acids result from beneficial shifts in the gut microbiome and may influence the inflammatory state of the skin.

Therefore, the study aims to investigate whether soy-derived isoflavone can reduce wrinkles and alter both gut microbiome and short-chain fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females, 50 to 70 years of age
* Fitzpatrick skin type I or II, based on skin melanin content
* BMI 18.5-35 kg/m2
* Must be willing to comply with all protocol requirements
* Must be willing to have flash photo facial images taken with the imaging systems

Exclusion Criteria:

* Any systemic or antibiotics (injected or oral) within 6 months of starting study
* Any topical antibiotic or benzoyl peroxide within 1 month of starting study or any subject unwilling to refrain from washout of topical antibacterial or benzoyl peroxide ingredient.
* Allergic to soy and milk products
* Fruit consumption > 2 cups/day
* Vegetable consumption > 3 cups/day for females
* Fruit juice consumption > 1 cup/day
* Coffee consumption > 1 cup per day
* Alcohol consumption ≥ 3 servings per week (1 serving = 1 bottle of beer, ½ glass of wine, or 1 shot of hard liquor)
* Self-reported malabsorption
* Any oral probiotic or prebiotic supplementation within past 1 month at the discretion of the investigator. Probiotic and prebiotic containing foods are NOT considered an exclusion.
* Subjects must have no history of malignancy or cancer or diagnosis of gastrointestinal inflammatory diseases, no history or diagnosis of epilepsy, no history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis)
* Has a condition or is on medication the investigator and/or designee believe could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results
* Is participating in a concurrent intervention based clinical research study
* Commencement of a new diet (such as the ketogenic diet) or supplements within the 1 month prior to initiating participation, at the discretion of the investigator.
* Use of medications that alter blood lipids, such as statins and anti-hyperlipidemic medications
* Is participating in or has participated in a intervention based facial study at this or any other facility in the past 2 weeks. Participation in survey-based studies are approved at the discretion of the investigator.
* Has a skin disease on face that will interfere with image collection and assessment in the opinion of the investigator
* Persons unwilling to avoid the following during the 4 weeks prior and during the duration of the study: self-tanning, spa tanning, sun tanning, or artificial tanning.
* Planned vacation to sunny destination with the intention of sun tanning during the duration of the study.
* Persons who regularly undergo sauna treatments (dry or wet) or who swim daily. Known allergy or irritation to the supplement or facial products utilized in the study
* Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco
* Prisoners
* Adults unable to consent
* Vegans and vegetarians

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Facial wrinkles | week 24
  Wrinkle severity score measured by Facial Image Analysis System

SECONDARY OUTCOMES:
Procollagen I expression | 24
  Assess with biopsy (optional participation)
Pigment intensity score | week 24
  Measured by the 3D Clarity Pro® Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA)
Blood levels of soy isoflavones and metabolites | week 24
  Blood samples will be collected
Gut microbiome | week 24
  Evaluate changes in the gut microbiome (Bifidobacteria and Lactobacilli, ratio of Firmicutes to Bacteroidetes) through stool samples
Blood lipidome | week 24
  Assess changes in butyrate, propionate, and acetate levels
Facial wrinkles | week 8
  Wrinkle score measured by Facial Image Analysis System
Facial wrinkles | week 16
  Wrinkle score measured by Facial Image Analysis System

IPD SHARING:
Plan to Share IPD: No